CLINICAL TRIAL: NCT07244380
Title: A Phase II Clinical Trial of S101 Autologous CAR-T Cell Injection for the Treatment of CD7-Positive Relapsed or Refractory T-Lymphoblastic Lymphoma/Leukemia (T-LBL/ALL).
Brief Title: Phase II Trial of S101 Autologous Anti-CD7 CAR-T Cells in Patients With R/R T-LBL/ALL.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARMA-II
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S101 CD7 CAR-T (Experimental): Autologous CD7-targeting CAR T cells, dosage 2*10^6/kg, intravenous injection once
  Interventions: Biological: Autologous CD7-targeting CAR T cells

INTERVENTIONS:
Biological: Autologous CD7-targeting CAR T cells — Autologous CD7-targeting CAR T cells, dosage 2*10^6/kg, intravenous injection once

SUMMARY:
To Evaluate the Efficacy and safety of S101 for Treating CD7-Positive Relapsed or Refractory T-LBL/ALL.

DETAILED DESCRIPTION:
This study is a Phase II, single-arm, open-label, single-infusion clinical trial designed to evaluate the clinical efficacy and safety of S101 in patients with CD7-positive relapsed or refractory T-lymphoblastic lymphoma/leukemia (T-LBL/ALL).

The primary objective： To evaluate the efficacy of S101 in patients with relapsed or refractory T-LBL/ALL.

The secondary objectives： To further characterize the efficacy, safety, pharmacokinetics and pharmacodynamics of S101 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 1.The subject or guardian must provide voluntary informed consent; 2.Heavily pretreated patients with relapsed or refractory T-LBL/ALL who lack effective therapeutic alternatives; 3.At screening, CD7 positivity of tumor cells must be documented by flow cytometry (on bone marrow or peripheral blood samples) and/or by immunohistochemistry (IHC) confirming CD7 expression on an extramedullary lesion biopsy; 4.If malignant cells are detected in the peripheral blood at screening, they must demonstrate a CD4-negative and CD8-negative (double-negative) immunophenotype as assessed by flow cytometry; 5.Male or female subjects, aged 18 to 75 years (inclusive); 6.Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2; 7.Estimated survival time>12 weeks.

Exclusion Criteria:

* 1.Patients with a history of allogeneic hematopoietic stem cell transplantation within the past 6 months are excluded; 2.Active or uncontrolled infection requiring systemic treatment at screening, excluding mild genitourinary and upper respiratory infections； 3.Participation in another clinical trial within 4 weeks prior to signing the informed consent form (ICF), OR the date of ICF signing occurring within 5 half-lives of the last dose from a previous investigational drug trial (whichever timeframe is longer); 4.Patients with previous treatment involving CAR-T cells or other gene-modified cell therapies are excluded; 5.Patients with acute GVHD (aGVHD) or moderate-to-severe chronic GVHD (cGVHD) within 4 weeks prior to screening, or those who have received systemic pharmacologic therapy for GVHD within 4 weeks prior to infusion; 6.Patients who have received extensive radiotherapy within 4 weeks prior to ICF signing, with the exception of non-target lesion radiotherapy administered for symptomatic palliation that may be permitted during the study period; 7.Women who are pregnant or lactating; 8.Any condition that, in the judgment of the Investigator, could increase the subject's risk or compromise the interpretation of the trial results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate after S101 infusion [Effectiveness] | 3 months
  Independent Review Committee (IRC)-assessed ORR at Month 3 post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Zhao, Principal Investigator — Peking University People's Hospital; Weili Zhao, Principal Investigator — Ruijin Hospital